CLINICAL TRIAL: NCT01247610
Title: Adult Outcome of Children With Attention-deficit/Hyperactivity Disorder
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Health Research Institutes, Taiwan (Other)
Responsible Party: Sponsor
Other Study IDs: 201003087R
Record Dates: First submitted 2010-11-22; First posted 2010-11-24 (Estimated); Last update posted 2021-09-05 (Actual); Status verified 2012-09

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — The subjects will receive blood withdrawal. The blood sample will be used for establishing lymphoblastoid cell lines, which will be used for molecular genetic experiments.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- ADHD group
- Control group

SUMMARY:
Attention deficit/hyperactivity disorder (ADHD) has been recognized as a common (5-8%), early-onset, long-term impairing, heterogeneous neuropsychiatric disorder with high heritability. Due to its lifelong impairments up to adulthood, adult ADHD has drawn much more attention in Western studies in the past decade; however, there has been no such study in Asian countries. The ultimate goals of this longitudinal follow-up study are to investigate the outcomes of a cohort of children with attention-deficit/hyperactivity (ADHD) and their healthy controls at young adulthood as the primary aim; and to test whether structural and functional brain connectivity can be endophenotypes of ADHD, to localize the brain area that are corresponding to methylphenidate treatment effects, and to identify the genetic variants corresponding to the persistence of ADHD, treatment effect of methylphenidate, neurocognitive dysfunction, and structural and functional dysconnectivity in the brain as the secondary aims. With the accomplishment of these goals, this study will provide the first-hand data on adult ADHD in non-western countries, and will be one of few world-class studies on the topics of neurocognitive and imaging genomics on adult ADHD.

DETAILED DESCRIPTION:
Primary specific aim:

To describe the manifestation and persistence of ADHD symptoms and to investigate the psychiatric, social, and executive functioning outcomes at young adulthood among children with ADHD;

Secondary specific aims

1. To identify early individual (clinical, behavioral, and executive functioning and other neurocognitive variables), family, school, environmental factors to predict the symptom persistence and a wide-range of outcomes at young adulthood;
2. To validate structural and functional connectivity of frontostriatal circuitry as imaging endophenotypes of ADHD by demonstrating that structural connectivity and functional connectivity of frontostriatal circuitry are altered in patients with ADHD and their unaffected siblings, are associated with ADHD symptoms, and are associated with genes related to dopamine neurotransmitter system;
3. To identify brain area that is corresponding to the effect of methylphenidate; and
4. To confirm reported candidate genes related to dopamine and noradrenergic neurotransmitter systems in the association with ADHD severity and subtypes (persistence, comorbidity, functional impairment, and treatment effects) and endophenotypes (executive function and structural and functional brain connectivity) such as DAT1, DRD4, MAO-A, ADRA2A, ADRA2C, NET, and COMT.

The sample consists of a cohort of 217 young adults (180 males, 83%) who were diagnosed of ADHD at childhood and 173 healthy controls (123 males, 71%). At their ages of 17-24 (around 6 years after their assessments at adolescence), they will receive psychiatric interviews (ADHD+SADS, CAADID) to make the diagnosis of ADHD and other psychiatric disorders and blood sample collection. They will complete the following questionnaires: ASRS and CAARS-S:S for adult ADHD symptoms, TPQ for personality characteristics, ASRI-4 for DSM-IV psychopathology, AAQoL and WFIRS for social functions, and PBI for parenting styles; and perform the WAIS-III for current IQ and Cambridge Neuropsychological Test Automated Batteries for attention control and executive functioning. Among the cohort subjects, 30 subjects with persistent ADHD and their same-sex and -handedness unaffected siblings (n = 30), 30 ADHD subjects who have DAT1 and/or good response to methylphenidate (repeated MRI assessment one week later) based on clinical assessment, and 30 subjects without lifetime ADHD and any psychiatric disorder will receive diffusion spectrum imaging (DSI) and resting state functional MRI assessments (total number of MRI assessments, 150). We will genotype 3'VNTR of DAT1 gene and other candidate genes involving dopaminergic and adrenergic systems (DRD4, MAO-A, ADRA2A, ADRA2C, NET, and COMT) for case-control association studies by using SNP and haplotype analysis.

We anticipate that this study (1) will provide the first prospective, longitudinal data of children with ADHD at late adolescence and young adulthood in Asian populations; (2) will be one of the first to establish a comprehensive, multi-dimensional dataset combining clinical, family, psychosocial, academic/vocational, neuropsychological, neuroimaging, and genetic data of young adults with ADHD. With the inclusion of imaging genetics data, the behavioral and neurocognitive phenotypes of ADHD can be validated, the imaging endophenotype can be tested, and image genetics approach may help identify genetic variants for ADHD.

ELIGIBILITY:
Inclusion Criteria:

1. Persistent ADHD combined type (Group 1, n=30): Subjects who have persistent diagnosis of ADHD, combined type, at adulthood according to the DSM-IV diagnostic criteria and who have same-sex unaffected siblings are included. If more than 30 subjects meet the inclusion criteria, the subjects with more severe ADHD symptoms based on the ASRS and K-SADS ratings will be included.
2. Unaffected sibling (Group 2, n=30): The same sex and handedness unaffected siblings of Group 1 will be recruited. They need to be re-assessed by psychiatric interview to confirm no lifetime diagnosis of ADHD.
3. Good response to MPH (Group 3, n=30): Subjects whose ADHD symptoms meet the DSM-IV symptom criteria at adulthood and who either have DAT1 genes (around 10% of Taiwanese children with ADHD15) or demonstrate good response to MPH based on clinical interview were recruited for offand on-stimulant DSI and resting state fMRI assessments.
4. Non-ADHD (Group 4, n=30): Among healthy controls without lifetime ADHD, the controls who do not have any lifetime psychiatric disorders and who do not have impaired neuropsychological function will be included. The control subjects will be matched for the age, gender, and handedness of Group 1.

Exclusion Criteria:

* These subjects will be excluded from the study if they have any of the following criteria: (1) Comorbidity with DSM-IV-TR diagnosis of pervasive developmental disorder, schizophrenia, schizoaffective disorder, delusional disorder, other psychotic disorder, organic psychosis, schizotypal personality disorder, bipolar disorder, depression, severe anxiety disorders or substance use; (2) With neurodegenerative disorder, epilepsy, involuntary movement disorder, congenital metabolic disorder, brain tumor, history of severe head trauma, and history of craniotomy; and (3)With visual or hearing impairments, or motor disability which may influence the process of MRI assessment. In addition, if the control subjects have ODD or CD, they will be excluded.

Ages: 17 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The sample will consist of (1) 217 adolescents (180 males, 83%) who were diagnosed of ADHD at childhood and followed up by Gau and consented to this follow-up study, and (2) 173 healthy controls (123, Males, 71%) without lifetime ADHD to late adolescence and adulthood. This cohort was established from 2005 to 2008. We will invite them for complete assessments 6 years after their assessments at adolescence according to the original assessment schedules from 2005-2008. The estimated age ranges are 17-24 years old.
Sampling Method: Non-Probability Sample
Enrollment: 390 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2015-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Shur-Fen Gau, MD, PhD, Principal Investigator — National Taiwan University Hospital & College of Medicine
Locations (1):
- National Taiwan Univeristy Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Chiang HL, Chen YJ, Lin HY, Tseng WI, Gau SS. Disorder-Specific Alteration in White Matter Structural Property in Adults With Autism Spectrum Disorder Relative to Adults With ADHD and Adult Controls. Hum Brain Mapp. 2017 Jan;38(1):384-395. doi: 10.1002/hbm.23367. Epub 2016 Sep 15. PMID 27630075